CLINICAL TRIAL: NCT05950178
Title: Validation of Apnea Test Conducted Using High-flow Oxygen Therapy in Patients With Clinical Brain Death
Brief Title: Validation of the Apnea Test Performed by High-flow Oxygen Therapy in Patients With Clinical Brain Death
Acronym: APNEAFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2022-10
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Brain Death
Keywords: Clinical brain death; Apnea test; High-flow oxygenation; Standard oxygen therapy; High-flow oxygen therapy
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled single-center trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical brain death (Other): The protocol is based on performing two consecutive apnea tests on a patient in clinical brain death in intensive care unit. The first apnea test will be conducted under standard oxygen therapy and confirms clinical brain death (standard procedure). The second apnea test (for the study) will be conducted under high-flow oxygen therapy. Only patients whose apnea test is initially validated under standard oxygen therapy will have the second apnea test under high-flow oxygen therapy.
  Interventions: Diagnostic Test: Apnea test under high-flow oxygenation

INTERVENTIONS:
Diagnostic Test: Apnea test under high-flow oxygenation — Apnea test under high-flow oxygenation in patients with a confirmed clinical brain death by a standard apnea test (under standard oxygen therapy)

SUMMARY:
Brain death is a clinical and paraclinical diagnosis established in a known etiological context. It involves the irreversible destruction of cerebral functions in a beating-heart individual.

In the context of organ and tissue donation from a critically ill patient, the clinical diagnosis of brain death is confirmed through a mandatory apnea test. This test is conducted by disconnecting the patient from the ventilator for a duration of 8 to 10 minutes. The test is considered validated when there is no spontaneous respiratory movement and the presence of hypercapnia. Hypercapnia is defined as a PaCO2 (carbon dioxide partial pressure) greater than 60 mmHg or an increase of more than 20 mmHg compared to the pre-ventilator disconnection capnia. These thresholds are meant to provide a strong stimulus to the respiratory centers, objectively confirming the absence of spontaneous ventilation.

In practice, the apnea test is performed under CPAP (Continuous Positive Airway Pressure) or by administering oxygen at 6-10L/min through the endotracheal tube.

High-flow oxygenation could be a simple alternative for the apnea test during the validation of the clinical diagnosis of brain death while reducing the risk of lung derecruitment and compromising organ viability and/or lung donation.

However, due to the high gas flow used (60 L/min), high-flow oxygenation can lead to a "washout" effect in the anatomical dead space, which may lower the carbon dioxide partial pressure. Consequently, even in a patient in a state of brain death, where spontaneous ventilation is absent by definition, it is not certain that the carbon dioxide partial pressure will increase to the threshold of 60 mmHg or more than 20 mmHg in 10 minutes during an apnea test conducted with high-flow oxygenation.

The purpose of this study is, therefore, to examine the feasibility of clinically diagnosing brain death through an apnea test performed with high-flow oxygenation.

To determine whether the validation criterion which involves observing an arterial capnia > 60 mmHg or an increase > 20 mmHg (compared to the capnia at the beginning of the test) after 10 minutes can be achieved during an apnea test conducted under high-flow oxygen therapy in patients with clinically confirmed brain death by standard apnea test (under standard oxygen therapy)

DETAILED DESCRIPTION:
The protocol is based on performing two consecutive apnea tests on a patient in clinical brain death in intensive care unit. The first apnea test will be conducted under standard oxygen therapy and confirms clinical brain death (standard procedure). The second apnea test (for the study) will be conducted under high-flow oxygen therapy. Only patients whose apnea test is initially validated under standard oxygen therapy will have the second apnea test under high-flow oxygen therapy.

After a standardized preoxygenation, the 1st apnea test will be performed under standard oxygen therapy through the endotracheal tube (flow at 8L/min) for 10 minutes. An arterial blood gas sampling will be sampled every 2 minutes during the1st apnea test.

The confirmation of clinical brain death by validating the apnea test under standard oxygen therapy will be done if the following two conditions are met: 1) absence of a spontaneous respiratory movements AND 2) an arterial capnia > 60 mmHg or an increase > 20 mmHg (compared to the capnia at the end of preoxygenation).

Then the patient will be reconnected to the ventilator for 15 minutes. A second standardized preoxygenation will be performed before the 2nd apnea test. The second apnea test will be performed under high-flow oxygen therapy through the endotracheal tube (flow at 50L/min, FiO2 100%) for 10 minutes. An arterial blood gas sampling will be sampled every 2 minutes during the1st apnea test.

Then the patient will be reconnected to the ventilator with the same settings before the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients in critical care with clinical brain death and potential organ and tissue donors for whom an apnea test is indicated.

Exclusion Criteria:

* Minor patients.
* Person under guardianship
* Protected Majors
* Not affiliated to French social security
* Pregnant women.
* Patients with a history of Chronic Obstructive Pulmonary Disease with a GOLD score of III or IV.
* Patients with at least one absolute contraindication to organ donation.
* Patients whose relatives have spontaneously expressed the patient's refusal to donate organs for therapeutic purposes.
* Patients on VA ECMO and, in general, any patient with a contraindication to performing the apnea test (DV, significant hemodynamic instability...).
* Patients whose relatives have refused the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients exceeding the hypercapnia threshold | 48 hours
  Percentage of patients exceeding the hypercapnia threshold after an apnea test conducted under high-flow oxygen therapy among patients who have already been validated for the apnea test under standard oxygen therapy.

SECONDARY OUTCOMES:
Time required after ventilator disconnection to exceed 60mmHg of PaCO2 or for which PaCO2 increases by more than 20mmHg compared to the PaCO2 before disconnection. | 48 hours
  Determine the maximum PaCO2 value reached by all included subjects at the 10-minute mark of the apnea test with high-flow oxygen therapy
Recording of PaO2 and PaCO2 values measured in 2-minute intervals during the standard apnea test and apnea test under high-flow oxygen therapy. | 48 hours
Recording of the PaO2/FiO2 ratio before and after each apnea test. | 48 hours
Recording of systolic blood pressure, measured every minute during the two apnea tests | 48 hours
  Describe the evolution of hemodynamic parameters during the standard apnea test and the apnea test with high-flow oxygen therapy
Recording of diastolic blood pressure, measured every minute during the two apnea tests | 48 hours
  Describe the evolution of hemodynamic parameters during the standard apnea test and the apnea test with high-flow oxygen therapy
Recording of heart rate,measured every minute during the two apnea tests | 48 hours
  Describe the evolution of hemodynamic parameters during the standard apnea test and the apnea test with high-flow oxygen therapy
Recording of pulse oximetry, measured every minute during the two apnea tests | 48 hours
  Describe the evolution of hemodynamic parameters during the standard apnea test and the apnea test with high-flow oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: Damien BARRIER, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR d'ORLEANS, Orléans, France

REFERENCES:
- [Background] Greer DM, Shemie SD, Lewis A, Torrance S, Varelas P, Goldenberg FD, Bernat JL, Souter M, Topcuoglu MA, Alexandrov AW, Baldisseri M, Bleck T, Citerio G, Dawson R, Hoppe A, Jacobe S, Manara A, Nakagawa TA, Pope TM, Silvester W, Thomson D, Al Rahma H, Badenes R, Baker AJ, Cerny V, Chang C, Chang TR, Gnedovskaya E, Han MK, Honeybul S, Jimenez E, Kuroda Y, Liu G, Mallick UK, Marquevich V, Mejia-Mantilla J, Piradov M, Quayyum S, Shrestha GS, Su YY, Timmons SD, Teitelbaum J, Videtta W, Zirpe K, Sung G. Determination of Brain Death/Death by Neurologic Criteria: The World Brain Death Project. JAMA. 2020 Sep 15;324(11):1078-1097. doi: 10.1001/jama.2020.11586. PMID 32761206
- [Background] Levesque S, Lessard MR, Nicole PC, Langevin S, LeBlanc F, Lauzier F, Brochu JG. Efficacy of a T-piece system and a continuous positive airway pressure system for apnea testing in the diagnosis of brain death. Crit Care Med. 2006 Aug;34(8):2213-6. doi: 10.1097/01.CCM.0000215114.46127.DA. PMID 16540953
- [Background] Lyons C, Callaghan M. Apnoeic oxygenation with high-flow nasal oxygen for laryngeal surgery: a case series. Anaesthesia. 2017 Nov;72(11):1379-1387. doi: 10.1111/anae.14036. PMID 29047136
- [Background] Fossat G, Nay MA, Jacquier S, Desmalles E, Boulain T. High-flow oxygen during spontaneous breathing trial for patients at high risk of weaning failure. Intensive Care Med. 2021 Aug;47(8):916-917. doi: 10.1007/s00134-021-06450-x. Epub 2021 Jun 14. No abstract available. PMID 34128122
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary. Am J Respir Crit Care Med. 2017 Mar 1;195(5):557-582. doi: 10.1164/rccm.201701-0218PP. PMID 28128970
- [Background] Wijdicks EF, Manno EM, Holets SR. Ventilator self-cycling may falsely suggest patient effort during brain death determination. Neurology. 2005 Sep 13;65(5):774. doi: 10.1212/01.wnl.0000174626.94197.62. No abstract available. PMID 16157923
- [Background] Shapiro BA. The apnea-PaCO2 relationship: some clinical and medico-legal considerations. J Clin Anesth. 1989;1(5):323-7. doi: 10.1016/0952-8180(89)90069-x. No abstract available. PMID 2516731
- [Background] Birks EJ, Burton PB, Owen VJ, Latif N, Nyawo B, Yacoub MH. Molecular and cellular mechanisms of donor heart dysfunction. Transplant Proc. 2001 Aug;33(5):2749-51. doi: 10.1016/s0041-1345(01)02178-9. No abstract available. PMID 11498147
- [Derived] Barrier D, Vanacker L, Muller G, Szychowiak P, Bretagnol A, Levebvre I, Narcisse E, Pascot L, Boulain T, Nay MA. Feasibility of High-Flow Oxygen Therapy in Apnea Testing for Brain Death Diagnosis. Crit Care Med. 2025 Jul 1;53(7):e1449-e1456. doi: 10.1097/CCM.0000000000006717. Epub 2025 May 19. PMID 40387463